CLINICAL TRIAL: NCT01190917
Title: Acute and Sustained Effects of Social Skills Intervention on Neural and Behavioral Outcomes in Children With ASD
Brief Title: Neural and Behavioral Outcomes of Social Skills Groups in Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO #09-0859; R21MH089236 (NIH)
Record Dates: First submitted 2010-08-20; First posted 2010-08-30 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder; Disorder; Autistic; Asperger Syndrome; social skills group; behavioral intervention; Imaging, Magnetic Resonance; fMRI; Functional MRI; MRI, Functional; Magnetic Resonance Imaging; Functional
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Disease; Asperger Syndrome | interventions — Cognitive Behavioral Therapy; Play Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy Group (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Social Play Group (Active Comparator)
  Interventions: Behavioral: Play Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The CBT social skills curriculum is manualized and anchored in CBT strategies, such as problem identification, affective education, performance feedback, and weekly homework activities to facilitate generalization. The curriculum is a compilation of lessons targeting key social deficits in children with ASD, such as nonverbal communication, emotion recognition, and theory of mind. Structured teaching includes defining skills, breaking them down into simple, concrete steps, modeling the skill through role-play, and introducing a game or activity to practice the target skill. The approach to the parent group will be psychoeducational with a focus on reviewing target skills, rationale for teaching target skills, homework, progress or obstacles, and identifying strategies to promote generalization. Parent information handouts will be provided.
  Arms: Cognitive Behavioral Therapy Group
Behavioral: Play Therapy — The social play group is manualized, led by a trained clinician and support staff, follows a specific routine, and contains a parent group component. Group leaders will follow participants' interests and suggestions for games. Group leaders utilize strategies such as reflective functioning statements on the child's behaviors to build emotion-focused play skills. The therapeutic setting incorporates play designed to encourage emotion-focused play including make-believe (dolls, houses), sensory (e.g. play-doh), and cooperative play (e.g. board games) toys. The approach to the parent group will be supportive rather than psychoeducational. Parents will set the agenda for discussion, facilitated by the group leader.
  Arms: Social Play Group

SUMMARY:
The purpose of this study is to compare two different treatment approaches to social skills groups for high-functioning children with Autism Spectrum Disorder (ASD). This project will examine changes in both behavior and the brain following treatment.

DETAILED DESCRIPTION:
Despite the fact that social skills impairments are the most persistent and pervasive symptoms affecting individuals with ASD, treatments targeting social skills have been the subject of few controlled investigations. The available literature suggests that cognitive behavioral techniques are commonly used and may improve targeted social skills in individuals with ASD. However, drawing firm conclusions about the efficacy of social skills treatment remains difficult, particularly with respect to maintenance of skills and generalization to natural settings, owing to methodological limitations of extant studies (e.g., small sample size, lack of manual-based curricula, minimal assessment of generalization or maintenance).

Several neuroimaging studies have found that individuals with ASD underactivate key brain regions involved in social cognition. However, there is also evidence to suggest that factors that increase attention to or interest in social stimuli are associated with more normal brain activity.

The purpose of this investigation is to examine the acute and sustained effects of social skills treatment on social cognition and the neural architecture that supports it. High-functioning children with ASD will be randomly assigned to a 12-week cognitive behavioral social skills group or a social play-based therapy group. For both types of groups, a parent session will be held concurrently. Functional MRI scans as well as behavioral assessments of social cognition, adaptive functioning, and symptom severity will be acquired at baseline, immediately following treatment, and at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 11 years of age
* Meets criteria for ASD according to psychiatric interview (DSM-IV), the Autism Diagnostic Observation Schedule-Generic, and the Autism Diagnostic Interview-Revised
* Verbal IQ ≥ 70, as measured by the Wechsler Intelligence Scale for Children-Fourth Edition or Wechsler Abbreviated Scale of Intelligence

Exclusion Criteria:

* History of psychiatric or neurological disorders other than ASD (e.g., schizophrenia, depression, seizure disorder)
* Within 30 days prior to the initial evaluation, beginning any new psychotropic medication or other therapeutic intervention (e.g., behavior, speech, physical/occupational, cognitive, nutritional therapy) that would confound the evaluation of the social skills groups
* Gross structural abnormality present in the brain (e.g., aneurysm)
* History of head trauma or loss of consciousness
* For any reason the child or parents appear unable to participate in study procedures

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Analysis of Nonverbal Accuracy-2* (DANVA2) | Week 0
  Assesses emotion recognition from facial expression, tone of voice, and posture. This instrument allows for the assessment of basic emotions conveyed by both adult and child models at high and low intensity. Nowicki and Carton [50] have shown that the DANVA2 has acceptable internal consistency for school age children and good test-retest reliability.
Diagnostic Analysis of Nonverbal Accuracy-2* (DANVA2) | Week 12
  Assesses emotion recognition from facial expression, tone of voice, and posture. This instrument allows for the assessment of basic emotions conveyed by both adult and child models at high and low intensity. Nowicki and Carton [50] have shown that the DANVA2 has acceptable internal consistency for school age children and good test-retest reliability.
Diagnostic Analysis of Nonverbal Accuracy-2* (DANVA2) | Week 24
  Assesses emotion recognition from facial expression, tone of voice, and posture. This instrument allows for the assessment of basic emotions conveyed by both adult and child models at high and low intensity. Nowicki and Carton [50] have shown that the DANVA2 has acceptable internal consistency for school age children and good test-retest reliability.
Reading the Mind in the Eyes Task - Child Version | Week 0
  The computerized children's version of the Eyes test is a reduced battery of 28-items measuring an individual's ability to interpret intentions and 'mentalizing' abilities, a hallmark social cognitive deficit in ASD. The adult RMET has shown sensitivity to change in clinical trials and the child version showed promising results in our preliminary analyses (see Preliminary Studies).
Reading the Mind in the Eyes Task - Child Version | Week 12
  The computerized children's version of the Eyes test is a reduced battery of 28-items measuring an individual's ability to interpret intentions and 'mentalizing' abilities, a hallmark social cognitive deficit in ASD. The adult RMET has shown sensitivity to change in clinical trials and the child version showed promising results in our preliminary analyses (see Preliminary Studies).
Reading the Mind in the Eyes Task - Child Version | Week 24
  The computerized children's version of the Eyes test is a reduced battery of 28-items measuring an individual's ability to interpret intentions and 'mentalizing' abilities, a hallmark social cognitive deficit in ASD. The adult RMET has shown sensitivity to change in clinical trials and the child version showed promising results in our preliminary analyses (see Preliminary Studies).
Functional Magnetic Resonance Imaging (fMRI) | Week 0
  We previously developed two activation tasks that tap different aspects of social cognition: 1) Interpreting Communicative Intent: Participants will view cartoon drawings of children while listening to short vignettes ending with a potentially ironic remark. Participants decide whether the speaker really meant what s/he said. 2) Affect and eye contact: Participants will view full-face pictures of people displaying happy, angry, fearful, or neutral affect. For each emotion, half of the faces show a direct gaze and half show a gaze aversion.
Functional Magnetic Resonance Imaging (fMRI) | Week 12
  We previously developed two activation tasks that tap different aspects of social cognition: 1) Interpreting Communicative Intent: Participants will view cartoon drawings of children while listening to short vignettes ending with a potentially ironic remark. Participants decide whether the speaker really meant what s/he said. 2) Affect and eye contact: Participants will view full-face pictures of people displaying happy, angry, fearful, or neutral affect. For each emotion, half of the faces show a direct gaze and half show a gaze aversion.
Functional Magnetic Resonance Imaging (fMRI) | Week 24
  We previously developed two activation tasks that tap different aspects of social cognition: 1) Interpreting Communicative Intent: Participants will view cartoon drawings of children while listening to short vignettes ending with a potentially ironic remark. Participants decide whether the speaker really meant what s/he said. 2) Affect and eye contact: Participants will view full-face pictures of people displaying happy, angry, fearful, or neutral affect. For each emotion, half of the faces show a direct gaze and half show a gaze aversion.

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | Week 0
  The SRS measures the severity of social impairment in natural settings, assessing social awareness, social information processing, reciprocal social communication, social anxiety/avoidance, and autistic preoccupations. This assessment will be completed by the child's parents and a classroom teacher, blind to intervention status, to reflect the opinion of more than one rater and allow for assessment of generalization across settings.
Social Responsiveness Scale (SRS) | Week 12
  The SRS measures the severity of social impairment in natural settings, assessing social awareness, social information processing, reciprocal social communication, social anxiety/avoidance, and autistic preoccupations. This assessment will be completed by the child's parents and a classroom teacher, blind to intervention status, to reflect the opinion of more than one rater and allow for assessment of generalization across settings.
Social Responsiveness Scale (SRS) | Week 24
  The SRS measures the severity of social impairment in natural settings, assessing social awareness, social information processing, reciprocal social communication, social anxiety/avoidance, and autistic preoccupations. This assessment will be completed by the child's parents and a classroom teacher, blind to intervention status, to reflect the opinion of more than one rater and allow for assessment of generalization across settings.
Strange Stories Task | Week 0
  These stories assess the ability to interpret nonliteral statements. Stories requiring the interpretation of a speaker's communicative intent will be read to participants. Questions probe whether the child understands that (a) a nonliteral statement has been made and (b) the intent behind the statement (i.e., was the speaker was lying, being sarcastic, joking?)
Strange Stories Task | Week 12
  These stories assess the ability to interpret nonliteral statements. Stories requiring the interpretation of a speaker's communicative intent will be read to participants. Questions probe whether the child understands that (a) a nonliteral statement has been made and (b) the intent behind the statement (i.e., was the speaker was lying, being sarcastic, joking?)
Strange Stories Task | Week 24
  These stories assess the ability to interpret nonliteral statements. Stories requiring the interpretation of a speaker's communicative intent will be read to participants. Questions probe whether the child understands that (a) a nonliteral statement has been made and (b) the intent behind the statement (i.e., was the speaker was lying, being sarcastic, joking?)
Vineland Adaptive Behavior Scales, Second Edition (Vineland II) | Week 0
  The Vineland II measures personal and social skills needed for everyday living. The Survey Form will be administered to the child's parents in a semi-structured interview format and the Teacher Checklist will be completed by a teacher blind to intervention status.
Vineland Adaptive Behavior Scales, Second Edition (Vineland II) | Week 12
  The Vineland II measures personal and social skills needed for everyday living. The Survey Form will be administered to the child's parents in a semi-structured interview format and the Teacher Checklist will be completed by a teacher blind to intervention status.
Autism Diagnostic Observation Schedule (ADOS) | Week 0
Autism Diagnostic Observation Schedule (ADOS) | Week 12
Direct Observation | 12 weeks (during treatment sessions)
  Structured direct observation procedures by blinded observers will be used to evaluate the following target behaviors: instrumental initiations, social initiations, response to initiations, and nonverbal behaviors. Direct observations will also be conducted during unstructured free-play sessions at baseline, mid-point, and endpoint.
Peer generalization assessment | Week 0
  An analogue play group will be used to evaluate generalization of treatment effects to unaffected, unfamiliar peers. The play group will consist of 4 children: 2 TD peers and 2 children with ASD (1 enrolled in CBT, 1 enrolled in social play). The analogue play session will consist of a 20-minute videotaped free-play period in which children are provided with cooperative play toys (e.g., make-believe, construction, and board games).
Peer generalization assessment | Week 12
  An analogue play group will be used to evaluate generalization of treatment effects to unaffected, unfamiliar peers. The play group will consist of 4 children: 2 TD peers and 2 children with ASD (1 enrolled in CBT, 1 enrolled in social play). The analogue play session will consist of a 20-minute videotaped free-play period in which children are provided with cooperative play toys (e.g., make-believe, construction, and board games).

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wang, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Latha Soorya, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine - Seaver Autism Center, New York, New York, United States

REFERENCES:
- [Derived] Soorya LV, Siper PM, Beck T, Soffes S, Halpern D, Gorenstein M, Kolevzon A, Buxbaum J, Wang AT. Randomized comparative trial of a social cognitive skills group for children with autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):208-216.e1. doi: 10.1016/j.jaac.2014.12.005. Epub 2014 Dec 20. PMID 25721186